CLINICAL TRIAL: NCT00939055
Title: A Randomized Controlled Trial of StomaphyX Versus Sham for Revisional Surgery in Post-Roux-en-Y Patients to Reduce Regained Weight
Brief Title: StomaphyX Versus Sham for Revisional Surgery in Post-Roux-en-Y Patients to Reduce Regained Weight
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on futility analysis, study would not meet primary endpoint.
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D00764
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- StomaphyX (Experimental): Post-Roux-en-Y revisional surgery using the StomaphyX device.
  Interventions: Device: StomaphyX
- Sham Procedure (Sham Comparator): No intervention
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Device: StomaphyX — Transoral incisionless fastening device that allows for GI tissue approximation and creation of full-thickness (serosa-to-serosa) plications.
  Other Names: transoral incisionless fastening device
  Arms: StomaphyX
Procedure: Sham procedure — False procedure
  Other Names: Placebo
  Arms: Sham Procedure

SUMMARY:
The Roux-en-Y gastric bypass (RNYGB) is a weight loss surgery that involves the creation of a small gastric pouch and rearrangement of the small intestine. Although RNYGB has been demonstrated as an effective bariatric procedure, a significant number of patients experience weight regain that is often associated with distended gastric anatomy. Open and laparoscopic approaches for revision are associated with higher complication rates than de novo procedures. This study will evaluate the safety and effectiveness of a revisional incisionless natural orifice surgery of the gastric pouch and stoma in producing weight loss in post-RNYGB patients who have experienced weight regain.

DETAILED DESCRIPTION:
The Roux-en-Y gastric bypass (RNYGB) is the most commonly performed bariatric procedure to treat morbid obesity 1. Numerous studies have documented the effectiveness of RNYGB in promoting excess weight loss (EWL) typically in the 65-80% range after 1.5 to 2 years 1. Despite the favorable short-term outcomes of this bariatric surgical procedure, approximately 10-40% of patients do not achieve successful long-term weight loss 2. The weight regain occurs typically within 2 to 7 years after RNYGB surgery and is associated primarily with dilation of the gastric pouch or stoma 3, 4. Several open and laparoscopic bariatric revision procedures have been used in an attempt to correct these dilations, but they all have been associated with serious complications such as perforations, obstruction, staple line disruption, blind loop syndrome, stoma ulcer, and incisional hernias 2, 5, 6. Because of this high rate of morbidity associated with revisional gastric bypass surgery, less invasive endoscopic procedures may become a preferred approach for weight regain after RNYGB 7, 8.

The StomaphyX delivery system with SerosaFuse fasteners consist of an ergonomic, flexible fastener delivery device and sterile polypropylene fastener implants. The unit is provided sterile and is a single use device. The polypropylene fasteners are proprietary and function only with the StomaphyX device. The device uses vacuum to invaginate tissue through a port into a chamber and fasten it using the H shaped polypropylene fasteners. The fastener delivery subsystem is comprised of 3 elements: stylet, pusher, and internal lumens. They run the length of the device, the pusher being a hollow tube that rides over the length of the stylet, both riding in the lumen. The stylet is sharp at the distal tip to pierce tissue. The fastener is loaded by snapping it onto the stylet in the loading port of the handle. When pushed by the operator, the stylet carries the fastener down the lumen which runs from the proximal handle assembly to the distal tissue port where it will eventually be deployed into the tissue. Durability of the SerosaFuse fasteners has been demonstrated during several clinical studies utilizing the EsophyX device 9-12.

Reason for Conducting the Present Study: The goal of this study was to investigate the safety and effectiveness of the StomaphyX device for revisional natural orifice surgery of the gastric pouch and gastrojejunostomy anastomosis (stoma) in RNYGB patients to reduce regained weight.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and less than 65 years of age
* BMI of at least 35 and no more than 40
* At least 2 years post-RNYGB surgery
* Initially achieved at least 60% EBL and a BMI 35 or less
* Regained at least 20% of pre-RNYGB excess weight at screening
* Stable weight or continued failure to lose weight for at least 3 months
* Enlarged gastric pouch (≥ 30 ml)
* Anatomy of upper GI judged suitable for revision using StomaphyX
* Completed successful nutritional screening
* Normal levels of vitamin D, iron/ferritin, calcium, and magnesium
* Absence of protein malnutrition confirmed by serum albumin > 3 g/dL
* Willing to cooperate with follow-up dietary recommendations and assessment tests
* Signed Informed Consent

Exclusion Criteria:

* Previous revisional bariatric surgery after RNYGB
* Esophageal stricture or any anatomic condition that precludes passage of the StomaphyX device to the gastric pouch
* Diabetes type I
* Causal factors for weight regain other than gastric pouch enlargement
* Serious complications experienced during and/or after RNYGB such as leaks, fistula, incisional hernia, ulcers, pulmonary embolism or deep venous thrombosis
* Pregnancy or plans of pregnancy in the next 12 months
* Immunosuppression
* ASA > 3
* Life expectancy less than one year
* An eating disorder, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Ed, Washington DC, American Psychiatric Association, 2000
* Active substance abuse
* Plans of smoking cessation in the next 12 months
* Treatment with weight-loss prescription drug therapy within three months preceding the screening
* Intention to use prescription drug therapy or the use of over-the-counter weight-loss preparations during the current study
* Current participant in another weight-loss study or other clinical trial
* Inflammatory bowel disease
* Presence of ulceration at the gastrojejunostomy anastomosis
* Portal hypertension
* Coagulation disorders or chronic use of anticoagulants
* Any active medical condition that would preclude the patient from completing the study or would result in an unreasonable risk to the patient

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita P. Courcoulas, MD MPH FACS, Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Eid GM, McCloskey CA, Eagleton JK, Lee LB, Courcoulas AP. StomaphyX vs a sham procedure for revisional surgery to reduce regained weight in Roux-en-Y gastric bypass patients : a randomized clinical trial. JAMA Surg. 2014 Apr;149(4):372-9. doi: 10.1001/jamasurg.2013.4051. PMID 24554030

RESULTS

PARTICIPANT FLOW:
Groups:
- StomaphyX: Post-Roux-en-Y revisional surgery using the StomaphyX device.
  StomaphyX: Revisional incisionless natural orifice surgery of gastric pouch and stoma.
  GI tissue approximation and creation of full-thickness (serosa-to-serosa) plications
Period: Overall Study
Arm/Group | StomaphyX | Sham Procedure
Started | 73 | 39
Completed | 69 | 39
Not Completed | 4 | 0
Not completed — Discontinuation prior to procedure | 4 | 0

BASELINE CHARACTERISTICS:
Population: A total of 112 patients entered the study. 73 patients were randomized to the treatment study arm while 39 patients were randomized to the control study arm. 4 patients discontinued participation prior to receiving the study procedure. Therefore, 108 patients were eligible for follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | StomaphyX | Sham Procedure | Total
Number analyzed (Participants) | 69 | 39 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (8.62) | 49 (7.35) | 49 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 35 | 102
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: A clinically significant reduction in pre-RNYGB excess weight, defined by ≥15% EBL and BMI < 35.
Time Frame: 12 month
Population: When futility analysis was performed, only 46 out of 108 patients had reached the 12 month primary endpoint. Analysis was performed on the 29 StomaphyX-treated patients to determine whether study objectives were met. Sham (control) patients were not analyzed.
Measure: Number; unit: participants
Groups:
- Sham: No intervention
Arm/Group | StomaphyX | Sham
Number analyzed (Participants) | 29 | 0
participants | 9 |

2. Secondary Outcome: Assessment of Changes to Quality of Life (QOL) Using a Validated QOL Questionnaire
Description: Quality of life as assessed by the Impact of Weight on Quality of Life Questionnaire (IWQOL-Lite); a ≥ 10 total score improvement from baseline (screening) will represent a clinically significant improvement.
Time Frame: 12 months
Population: Secondary endpoint was not analyzed.
Arm/Group | StomaphyX | Sham Procedure
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the 12-month post-op visit for treatment and sham patients. The blind was broken for all patients due to premature termination of the study.
Description: 112 subjects enrolled/randomized:73 StomaphyX, 39 Sham. 108 treated:69 StomaphyX, 39 Sham. 112 patients were considered at risk for all cause mortality; 108 (69 StomaphyX, 39 Sham) considered at risk for serious/other adverse events. The 4 patients not included were in StomaphyX arm: 2 withdrawn prior to treatment at investigator discretion. Surgery was aborted on the other 2; treatment not completed as device couldn't be inserted. These 4 followed per site standard of care, outside study.
Arm/Group | StomaphyX | Sham
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/39
Serious Adverse Events (participants affected / at risk) | 3/69 | 0/39
Other Adverse Events (participants affected / at risk) | 18/69 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StomaphyX (N=69) | Sham (N=39)
Perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Small perforation in posterior gastrojejunostomy anastomosis.
Tachycardia, Infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StomaphyX (N=69) | Sham (N=39)
Nausea (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Sore Neck (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Temporary epigastric or abdominal pain (Injury, poisoning and procedural complications) | 11 (11) | 1 (1) — can be treated with standard pain medication
Pharyngolaryngeal pain (e.g. throat pain) (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Burps a lot after eating (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Temporary dysphagia (i.e. difficulty swallowing) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — due to swelling

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No